CLINICAL TRIAL: NCT02015923
Title: Multicenter Randomized Study in Patients With Colorectal Cancer With Unresectable Metastases. Impact of Resection vs no Resection of the Primary Tumour as a Survival Factor
Brief Title: Resection vs no Resection of the Primary in Colorectal Cancer With Unresectable Metastases
Acronym: CCRe-IV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties surrounding recruiting patients
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Sebastiano Biondo, Phd, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01CCRe-IV; 2013-001688-22 (EudraCT Number)
Record Dates: First submitted 2013-11-28; First posted 2013-12-19 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Colonic Cancer; Unresectable Metastasis Originating in Colonic Cancer
Keywords: Colonic cancer; Metastasis
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis | interventions — Folfox protocol; IFL protocol; FOLFOXIRI protocol; Bevacizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colonic resection (Experimental): Arm A (experimental): surgery (complete tumoral resection; R0) followed by chemotherapy, regimen according to each center.
  Interventions: Procedure: Colonic resection; Drug: Chemotherapy- scheme
- Chemotherapy (Active Comparator): Arm B (control): chemotherapy alone, regimen according to each center
  Interventions: Procedure: Colonic resection; Drug: Chemotherapy- scheme

INTERVENTIONS:
Procedure: Colonic resection — Colonic cancer resection, R0 No surgical intervention on metastasis
Drug: Chemotherapy- scheme — Chemotherapy, specified in each center with or without biological drugs
  Other Names: FOLFOX-4; FOLFOX-6; FOLFIRI; FOLFOXIRI; CAPOX; CETUXIMAX / BEVACIZUMAB/PANITUMUMAB

SUMMARY:
Main outcome: Assess the impact of cancer-related survival at 2 years in patients with unresectable metastatic colorectal cancer treated with chemotherapy alone versus surgery followed by chemotherapy. To assess overall survival. To evaluate postoperative morbidity and mortality in patients treated with resection of the primary tumor. Assess complications and meed for surgery in patients treated with systemic chemotherapy only during the course of the disease. Identify and describe the complications related to chemotherapy and toxicity in the short and medium term systemic treatment. Assessing the quality of life questionnaire QLQ-C30 and QLQ-CR29. To study prognostic survival factors.

Method: multicenter randomized clinical trail (22 hospitals). Two parallel group in which to evaluate two therapeutic strategies for colorectal cancer metastasis unresectable stage IV: chemotherapy alone versus primary tumor resection plus chemotherapy.

Subjects: patients with unresectable nonmetastatic colorectal cancer. Hypothesis:Surgical resection of the primary tumor in stage IV colorectal patients with unresectable synchronous metastases increases by 14% overall survival compared to patients receiving systemic treatment with chemotherapy without resection of the primary tumor (survival of 34% vs 20%).

DETAILED DESCRIPTION:
Intervention: Arm B (control): chemotherapy alone, regimen according to each center. Arm A (experimental): surgery (complete tumoral resection; R0) followed by chemotherapy, regimen according to each center. Statistical Analysis: A power analysis showed that to assure a significance level of 0,05 and a beta error 0.20. 168 patients are necessary in each arm. It has been estimated a loss rate of up to 10%.

Differences between groups will be analyzed by t, U, X2, exact test and survival will be assessed according to Kaplan and Meier method. Evaluation of safety of the trial will be made in the middle of the study statistically

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer above to 12 cm from the anal verge
* unresectable synchronous metastases
* no contraindications for chemotherapy
* absence of peritoneal carcinomatosis, central nervous system o bone metastasis.
* performance status ECOG ≤ 2 (Eastern Cooperative Oncology Group)
* uncontrolled concomitant medical conditions that may compromise to chemotherapy
* significant symptomatic cardiac disease
* not pregnancy or breastfeeding

Exclusion Criteria:

* Cases of rectal tumours below 12cm from anal verge, or locally advanced tumours invading blood vessels, nerves or bone.
* Multiple bone metastasis or central nervous system metastasis
* Other neoplastic disease in the 5 previous years, except squamous or basal cell skin carcinoma or cervical "in situ" carcinoma
* Significant heart disease (chronic congestive heart failure, symptomatic coronary disease) or myocardial infarction in the previous 6 months
* Peripheral neuropathy
* Patients who do not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-12; Primary Completion 2019-06 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Assess the impact of overall survival in patients with unresectable metastatic colorectal cancer treated with chemotherapy alone vs surgery followed by chemotherapy. | up to 2 years
  The percentage of patients who are still alive for follow-up at 2 years after randomization.

SECONDARY OUTCOMES:
Postoperative morbidity and mortality. | 30 days postoperatively
  Postoperative complications were classified according to the Dindo-Clavien classification.
  Mortality within 30 days after surgery
Complications in patients treated with systemic chemotherapy | up to 2 years
  The toxicity will be evaluated and documented according to the CTCAE version 4.0.
Questionnaire Quality of life CR29 | up to 2 years
  Specific questionnaire for colon cancer
Study of possible survival factors | up to 2 years
  Identify factors that may influence patient survival before applying any treatment (demographics, clinicals and analitycal factors, tumor characteristics; ...)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, Sponsor, Study Chair — Hospital Universitari de Bellvitge; Javier Vaqué, Principal Investigator — Hospital Universitario La Fe; Juan García Armengol, Principal Investigator — Hospital General Universitario de Valencia; Laura Mora, Principal Investigator — Corporacion Parc Tauli; Ignasi Camps Ausàs, Principal Investigator — Hospital Universitari Gemans Tiras i Pujol; Miguel Pera Román, Principal Investigator — Hospital Univesitari del Mar; Eduardo Targarona Soler, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Lorenzo Viso Pons, Principal Investigator — Hospital de Sant Joan Despí Moisès Broggi; José Manuel Ramírez Rodríguez, Principal Investigator — Hospital Clínico Univeristario "Lozano Blesa"; David Julià Bergkvist, Principal Investigator — Hospital Universitari de Girona DrJosep Trueta; Teresa García Martínez, Principal Investigator — Complejo Hospitalario Universitario de Vigo; Mario Álvarez Gallego, Principal Investigator — Hospital Univerisitario La Paz; José María Enríquez Navascués, Principal Investigator — Hospital Donostia; Fernando de la Portilla de Juan, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Miguel Angel Ciga, Principal Investigator — Complejo Hospitalario de Navarra; Eloy Espín Basany, Principal Investigator — hospital Universitari de la Vall D'Hebron; Manuel Ferrer Márquez, Principal Investigator — Complejo Hospitalario Torrecárdenas; Jesús Abrisqueta Carrión, Principal Investigator — Hospital Universitario Virgen de la Arrixaca; José Errasti Alustiza, Principal Investigator — Hospital Universitario Araba; Alberto Parajó Calvo, Principal Investigator — Complejo Hospitalario Universitario de Orense; Carlos Moreno Sanz, Principal Investigator — Complejo Hospitalario La Mancha Centro; Alejando Espí Macías, Principal Investigator — Hospital Clínico Universitario de Valencia; Ricard Frago Montanuy, Principal Investigator — Hospital Universitari de Bellvitge
Locations (22):
- Spain (22):
  - Hospital Universitario Araba, Vitoria-Gasteiz, Araba
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Complejo Hospitalario La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Univesitari Vall d'Hebron, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitari de Girona DrJosep Trueta, Girona
  - Hospital Univerisitario La Paz, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Universitari i Politècnic la Fe, Valencia
  - Hospital Clínico Univeristario "Lozano Blesa", Zaragoza

REFERENCES:
- [Derived] Rahbari NN, Biondo S, Frago R, Feisst M, Kreisler E, Rossion I, Serrano M, Jager D, Lehmann M, Sommer F, Dignass A, Bolling C, Vogel I, Bork U, Buchler MW, Folprecht G, Kieser M, Lordick F, Weitz J; SYNCHRONOUS and CCRe-IV Trial Groups. Primary Tumor Resection Before Systemic Therapy in Patients With Colon Cancer and Unresectable Metastases: Combined Results of the SYNCHRONOUS and CCRe-IV Trials. J Clin Oncol. 2024 May 1;42(13):1531-1541. doi: 10.1200/JCO.23.01540. Epub 2024 Feb 27. PMID 38412408
- [Derived] Biondo S, Frago R, Kreisler E, Espin-Basany E; Spanish CR4 Group. Impact of resection versus no resection of the primary tumor on survival in patients with colorectal cancer and synchronous unresectable metastases: protocol for a randomized multicenter study (CR4). Int J Colorectal Dis. 2017 Jul;32(7):1085-1090. doi: 10.1007/s00384-017-2827-3. Epub 2017 May 11. PMID 28497402